CLINICAL TRIAL: NCT06778629
Title: Evaluation of the Effectiveness of Transversalis Fascia Plane Block in Patients Undergoing Laparoscopic Inguinal Hernia Repair
Brief Title: Transversalis Fascia Plane Block for Laparoscopic Inguinal Hernia Repair
Acronym: TFPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ayse Ince, Assist Prof, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 5
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Laparoscopic Inguinal Hernia Repair; Acute Post Operative Pain
Keywords: Transversalis Fascia Plane Block; Acute Postoperative Pain; Laparoscopic Inguinal Hernia Repair
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 with American Society of Anesthesiologists (ASA) classification I-II scheduled for laparoscopic inguinal hernia repair operation will be included in the study. Before entering the operating room, patients will be randomly divided into two groups (Group T = TFPB group, Group K = control group), each with 30 patients.
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcomes assessor and participants will be blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T = TFPB group (Experimental): Transversalis Fascia Plane block will be performed. Local anesthetic infiltration to port entrance sites at the beginning of the operation and standard postoperative pain management protocols will be applied.
  Interventions: Procedure: Transversalis Fascia Plane Block; Procedure: Post Operative Pain Management; Procedure: Port Site Infiltration
- Group K = Control group (Active Comparator): Local anesthetic infiltration to port entrance sites at the beginning of the operation and standard postoperative pain management protocols will be applied. No plane block will be applied.
  Interventions: Procedure: Post Operative Pain Management; Procedure: Port Site Infiltration

INTERVENTIONS:
Procedure: Transversalis Fascia Plane Block — After the wound closure is completed and the patient is still under general anesthesia the TFPB will be performed. As the patient is in the supine position, the high-frequency linear US probe (11-12 MHz, Vivid Q) and a 22-G 80-mm needle (Stimuplex® Ultra 360®, Braun, USA) will be placed longitudinally, 2-3 cm laterally, just above the iliac crest at the mid-axillary line. After the external oblique, internal oblique, and transversus abdominis muscles are distinguished, the common aponeurosis of the transversus abdominis and the internal oblique muscle will be found. The block needle will be directed from anterior to posterior, using an in-plane technique, the block needle will be advanced and the block location will be confirmed by injecting 5 ml of saline. Once the block location is confirmed, 30 ml of 0.25% bupivacaine (Buvicaine, Polifarma ®) will be applied between the transversus abdominis muscle and transversalis fascia.
  Arms: Group T = TFPB group
Procedure: Post Operative Pain Management — Acetaminophen 1 gr (Paracerol, Polifarma®) intravenous (IV), and tramadol (Contramal, Abdi İbrahim®) 100 mg IV will be administered to all patients 30 minutes before wound closure. After surgery, Acetaminophen (Paracerol, Polifarma®) 1 gr IV, and tramadol (Contramal, Abdi İbrahim®) 100 mg IV will be given three times a day. Another anesthesiologist will assess patients after surgery. If the patient's pain score (NRS) is 4 or higher, IV pethidine (Aldolan, Liba Laboratory ®) 0,5 mg/kg will be given as a rescue analgesic.
Procedure: Port Site Infiltration — A total of 20 ml of 0.25% bupivacaine ( (Buvicaine, Polifarma ®) will be applied to the trocar entry points by the surgeon at the beginning of the operation, before entering the trocars.

SUMMARY:
Transversalis Fascia Plane Block (TFPB) is a trunk block that blocks the T12- L2 spinal nerves by injection of local anesthetic between the transversus abdominis muscle and transversalis fascia on the lateral abdominal wall. The block's positive effects on postoperative analgesia have been shown in many abdominal surgeries, including open-technique inguinal hernia repair.

This study aimed to investigate the effectiveness of ultrasound (US) guided TFPB on postoperative pain control for postoperative analgesia management after laparoscopic inguinal hernia repair.

DETAILED DESCRIPTION:
Inguinal hernia repairs are one of the most common general surgical operations and are generally performed with laparoscopic technique. Even laparoscopic inguinal hernia repair results in less acute postoperative pain compared to the open technique, untreated early pain may prolong hospital stay, exacerbate general discomfort, and affect the length of recovery, which may also have social and -economic implications. Opioids, due to their potent analgesic effects are used as a component of multimodal analgesia in the postoperative period. Despite their advantages, opioids may be related to pulmonary complications, postoperative delayed recovery due to ileus, nausea, and vomiting; and prolonged hospital stay. The use of interfascial plane blocks for pain management has increased recently, as ultrasonography (USG) has become a part of daily routine. Interfascial plane blocks provide effective postoperative analgesia.

Transversalis Fascia Plane Block (TFPB) is a body block that blocks the T12-L2 spinal nerves by injection of local anesthetic between the transversus abdominis muscle and transversalis fascia on the lateral abdominal wall Its positive effects on postoperative analgesia have been shown in many abdominal surgeries, including open technique inguinal hernia repair.

This study aimed to investigate the effectiveness of ultrasound (US) guided TFPB on postoperative pain control for postoperative analgesia management after laparoscopic inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I- II Patients
* Unilateral Inguinal Hernia Repair Surgery
* Elective Operations

Exclusion Criteria:

* Patients with a history of chronic pain
* Evidence of infection in the intervention area
* Allergy to local anesthetics
* Coagulopathy
* Body-mass index (BMI) ≥ 30
* Body weight ≤ 50 kg
* Patients who do not agree to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Rescue analgesic use | Need for rescue analgesics at 1, 3, 6, 12,18, and 24 hours postoperatively.
  The primary aim is to compare the rescue analgesia amount and its time used in the postoperative 24-hour period

SECONDARY OUTCOMES:
Compare postoperative pain scores (NRS scores) | NRS scores at rest and while moving will be evaluated and recorded at 1, 3, 6, 12,18, and 24 hours postoperatively.
  The secondary aim is to compare the pain scores at rest and with movement. Postoperative pain assessment will be performed using the Numerical Rating Scale (NRS) (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded. Low NRS is associated with better pain control.
Side effects and complications | Side effects and complications will be evaluated and recorded at 1, 3, 6, 12,18, and 24 hours postoperatively
  To evaluate block-related complications and side effects (allergic reaction, nausea, vomiting)- block or opioid related

CONTACTS AND LOCATIONS:
Overall Officials: BAHADIR CIFTCI, Study Chair — ISTANBUL MUH
Locations (1):
- Istanbul Medipol University Mega Hospital Complex, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data (IPD).

REFERENCES:
- [Result] Celik HK, Tulgar S, Buk OF, Koc K, Unal M, Genc C, Suren M. Comparison of the analgesic efficacy of the ultrasound-guided transversalis fascia plane block and erector spinae plane block in patients undergoing open inguinal hernia repair under spinal anesthesia. Korean J Anesthesiol. 2024 Apr;77(2):255-264. doi: 10.4097/kja.23404. Epub 2024 Jan 8. PMID 38185619
- [Result] Pinarbasi A, Altiparmak B, Korkmaz Toker M, Pirincci F, Ugur B. Ultrasound-guided transversalis fascia plane block or transversus abdominis plane block for recovery after caesarean section: A randomised clinical trial. Eur J Anaesthesiol. 2024 Oct 1;41(10):769-778. doi: 10.1097/EJA.0000000000002041. Epub 2024 Jul 22. PMID 39039833
- [Result] Hebbard PD. Transversalis fascia plane block, a novel ultrasound-guided abdominal wall nerve block. Can J Anaesth. 2009 Aug;56(8):618-20. doi: 10.1007/s12630-009-9110-1. Epub 2009 Jun 4. No abstract available. PMID 19495909
- [Result] Xu LS, Li Q, Wang Y, Wang JW, Wang S, Wu CW, Cao TT, Xia YB, Huang XX, Xu L. Current status and progress of laparoscopic inguinal hernia repair: A review. Medicine (Baltimore). 2023 Aug 4;102(31):e34554. doi: 10.1097/MD.0000000000034554. PMID 37543778
- [Result] Tolver MA, Rosenberg J, Bisgaard T. Early pain after laparoscopic inguinal hernia repair. A qualitative systematic review. Acta Anaesthesiol Scand. 2012 May;56(5):549-57. doi: 10.1111/j.1399-6576.2011.02633.x. Epub 2012 Jan 19. PMID 22260427